CLINICAL TRIAL: NCT02179372
Title: Modulation of Fecal Calprotectin by Eicosapentaenoic Free Fatty Acid in Inflammatory Bowel Diseases
Brief Title: Eicosapentaenoic Free Fatty Acid and Fecal Calprotectin in Inflammatory Bowel Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, andrea belluzzi, MD phD, Consultant in Gastroenterology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPA/CALPRO
Record Dates: First submitted 2014-06-29; First posted 2014-07-01 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eicosapentaenoic acid (Experimental): Subject with Cronn's Disease and/or Ulcerative colitis in clinical remission will receive 2 g/day of eicosapentaenoic acid for 6 months
  Interventions: Dietary Supplement: Eicosapentaenoic acid
- Medium chain fatty acid (placebo) (Placebo Comparator): Subjects with Crohn's Disease and/or Ulcerative colitis will be receive 2 g/day of medium chain fatty acid for 6 months
  Interventions: Dietary Supplement: Medium chain fatty acid (placebo)

INTERVENTIONS:
Dietary Supplement: Eicosapentaenoic acid — 30 subject with Crohn's Disease and/or Ulcerative Colitis in clinical remission but with fecal calprotectin value >150 μg/g will recive 2 g/day of Eicosapentaenoic acid for 6 months treatment. At 3 months and 6 months, fecal calprotectin and clinical activity (CDAI for Crohn's Disease and SCCAI for Ulcerative Colitis) will be measured. The effect of Eicosapentaenoic acid on fecal calprotectin level will be monitored. Clinical relapses will be considered during the study.
  Other Names: ALFA TM (S.L.A. Pharma A.G. Switzerland)
  Arms: Eicosapentaenoic acid
Dietary Supplement: Medium chain fatty acid (placebo) — 30 subject with Crohn's Disease and/or Ulcerative Colitis in clinical remission but with fecal calprotectin value >150 μg/g will recive 2 g/day of medium chain fatty acids for 6 months treatment. At 3 months and 6 months, fecal calprotectin and clinical activity (CDAI for Crohn's Disease and SCCAI for Ulcerative Colitis) will be measured.
  Arms: Medium chain fatty acid (placebo)

SUMMARY:
The aim of this study is to test Eicosapentaenoic free fatty acid's effects on calprotectin levels in IBD patients in clinical remission. During the study fecal calprotectin levels will be measured every 3 months and clinical flares will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged between18 and 80 years.
* Patients with Ulcerative Colitis (diagnosed on the base of clinic, endoscopic and histologic criteria) in clinical remission (SCCAI = 0) from at least 3 months and in stable therapy (without therapeutic modifications in the three previous months) with 5-ASA, immunomodulators and/or biologics.
* Patients affected by Crohn's Disease (diagnosed on the base of clinic, endoscopic and histologic criteria) ) in clinical remission (CDAI < 150) from at least 3 months and in stable therapy (without therapeutic modifications in the three previous months) with 5-ASA, immunomodulators and/or biologics.
* Fecal calprotectin at baseline > 150 μg/g.

Exclusion Criteria:

* Patients affected by Ulcerative Colitis and Crohn's Disease respectively with a SCCAI ≥ 1 and a CDAI ≥150.
* Patients on steroid therapy.
* Patients in therapy wih warfarin or other anticoagulants.
* Known or supposed ipersensitivity to eicosapentaenoic acid/omega 3.
* Women in fertile age which refuse to use contracceptives specified in the study (oral contraception, IUD) and breastfeed women.
* Patients with severe clinical conditions which the investigator consider to controindicate patient partecipation at the study.
* Therapy modifications and/or assumption of sperimental therapies within three months before the study inclusion.
* Patients unable to follow protocol procedures and to sign the informate consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
changes in fecal calprotectin levels | baseline, 3 months and at 6 months

SECONDARY OUTCOMES:
number of clinical flares of diseases | at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico Sant'Orsola Malpighi, Bologna, Bologna, Italy

REFERENCES:
- [Derived] Scaioli E, Sartini A, Bellanova M, Campieri M, Festi D, Bazzoli F, Belluzzi A. Eicosapentaenoic Acid Reduces Fecal Levels of Calprotectin and Prevents Relapse in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1268-1275.e2. doi: 10.1016/j.cgh.2018.01.036. Epub 2018 Jan 31. PMID 29391271